CLINICAL TRIAL: NCT06068686
Title: Effect of Vildagliptin Versus Glimepiride on Copeptin and Fetuin-A in Type 2 Diabetic Patients
Brief Title: Vildagliptin Versus Glimepiride in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vilda. vs Glim. in T2D
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; glimepiride; Tablets

STUDY DESIGN:
Intervention Model Description: 70 enrolled patients will be divided into two groups (35 each); both groups will be patients who are uncontrolled and already on metformin, group I will receive vildagliptin as an add-on therapy while group II will receive glimepiride.
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vildagliptin (Experimental): Group I (N=35) are patients who the endocrinologist prescribed them Vildagliptin 50mg /tab plus their Metformin 500mg /tab once daily for 12 weeks to control their blood sugar level.
  Interventions: Drug: Vildagliptin 50 MG
- Glimepiride (Active Comparator): Group II (N=35) are patients who the endocrinologist prescribed them Glimepiride 3mg / tab plus Metformin 500mg /tab once daily for 12 weeks.
  Interventions: Drug: Glimepiride 3 Mg Oral Tablet

INTERVENTIONS:
Drug: Vildagliptin 50 MG — vildagliptin plus their metformin.
  Other Names: Vildagliptin
  Arms: Vildagliptin
Drug: Glimepiride 3 Mg Oral Tablet — glimepiride plus their metformin
  Other Names: Amaryl
  Arms: Glimepiride

SUMMARY:
The aim of this study is to evaluate the effect of vildagliptin on copeptin in comparison to glimepiride, and whether copeptin could be used as a marker for the efficacy of vildagliptin in type 2 diabetes mellitus patients, and how copeptin correlates with other diabetic and cardiac markers.

DETAILED DESCRIPTION:
1. Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University.
2. All participants agreed to take part in this clinical study and provide informed consent.
3. Patients with uncontrolled DM type 2 who are on metformin will be enrolled from endocrinology clinic at Damanhour general hospital.
4. Serum samples will be collected for measuring the biomarkers.
5. All enrolled patients will be divided into two groups; both groups will be patients who are uncontrolled and already on metformin, group I will receive vildagliptin as an add-on therapy while group II will receive glimepiride.
6. All patients will be followed up during 12 week period.
7. At the end of the 12 week period, serum samples will be recollected for measuring the biomarkers after treatment.
8. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
9. Measuring outcome: The primary outcome is the change of serum levels of the measured markers after 12 weeks.
10. Results, conclusion, discussion and recommendations will be given. Methodology

    * Copeptin and NT-proBNP will be determined by ELISA.
    * Lipid profile will be measured.
    * Fasting blood glucose and Insulin will be measured and HOMA-IR will be calculated for all subjects.
    * Body weight and blood pressure will be measured.
    * HbA1C will be measured.

ELIGIBILITY:
Inclusion criteria

• 70 uncontrolled adult patients with Type II-diabetes mellitus

Exclusion criteria

* Hepatic impairment.
* Active malignancy.
* Planned surgical intervention.
* Any signs of hypersensitivity or contraindication to study drugs developed.
* Addition of any anti-diabetic medications or insulin during follows up.
* Chronic inflammatory disease (i.e. inflammatory bowel disease, lupus, inflammatory arthritis, rheumatoid arthritis) or chronic infection (i.e. chronic diabetic foot infection).
* Pregnancy, lactation or child-bearing potential.
* Cardiac disease.
* Renal impairment.
* History of T1DM, SIAD, or diabetes insipidus.
* Therapy with any diuretic or a medication affecting the RAAS.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Copeptin Concentration (pg/ml) | 3 month
  Copeptin serum Level
NT-proBNP Concentration (pg/ml) | 3 Months
  NT-proBNP serum Level

SECONDARY OUTCOMES:
Fasting blood glucose (mg/dl) | 3 month
  Fasting Blood Glucose level

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass Prof., Study Chair — Damanhour University
Locations (1):
- Damanhour Teaching Hospital, General Organization for Teaching Hospitals and Institutes., Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No